CLINICAL TRIAL: NCT04858841
Title: The Primary Prevention Study of Post-Ischemic Stroke Epilepsy
Brief Title: Post-stroke Epilepsy: Primary Prophylaxis Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chin-Wei Huang, Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A-BR-108-107
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Middle Cerebral Artery Stroke
MeSH Terms: conditions — Infarction, Middle Cerebral Artery | interventions — Levetiracetam; perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Levetiracetam (Experimental): The group receives oral levetiracetam.
  Interventions: Drug: Levetiracetam Oral Product
- Perampanel (Experimental): The group receives oral perampanel.
  Interventions: Drug: Perampanel Oral Product
- Placebo (Placebo Comparator): The group receives oral placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam Oral Product — Administer levetiracetam powder once a day in eligible patients
  Other Names: keppra
  Arms: Levetiracetam
Drug: Perampanel Oral Product — Administer perampanel powder once a day in eligible patients
  Other Names: fycompa
  Arms: Perampanel
Drug: Placebo — Administer placebo powder once a day in eligible patients
  Arms: Placebo

SUMMARY:
Advance in stroke treatment have resulted in a dramatic reduction in the stroke mortality, however, the number of stroke survivors living with morbidity has increased significantly. As we know, post-stroke epilepsy has been identified as a significant clinical issue in stroke survivors and stroke is the most common cause of epilepsy in older adults and for patients aged more than 65, post-stroke epilepsy accounts for 30-50% of new-onset seizures. Our previous study documented seizures during stroke presentation and during hospitalization would worsen the overall morbidity and mortality, suggesting the importance of awareness in seizure care in acute ischemic stroke.

As current studies only focus on anti-seizure/anti-convulsion after the appearance of late-onset seizures, without the intervention of the epileptogenesis, it is important to develop a potential novel prophylactic treatment on patients with acute severe stroke to prevent from late occurrence of seizures and epilepsy.

We have previously done researches on the medications that might have potential of anti-epileptogenesis in pilocarpine-induced animal models, supporting the concept of antiepileptogenesis, giving intervention immediately following a brain insult.

The results of some earlier anecdotal reports or small studies on prophylactic use of antiepileptic drug (AED) therapy in stroke, either hemorrhagic or ischemic strokes, remain inconclusive. There still lacks a well-established case-control study on prophylaxis of post-stroke epilepsy, with the early intervention of AED therapy with potential of anti-epileptogenesis in the phase of epileptogenesis.

Based on our clinical experience, and laboratory researches, we have noted two non-conventional AEDs, levetiracetam (LEV) and perampanel (PER) with potential of anti-epileptogenesis. It is justified to evaluate if early administration of LEV or PER in patients with acute major stroke as a prophylactic therapy could hamper the development of epileptogenesis and the later post-stroke epilepsy.

We aim to conduct a randomized case-control study to evaluate if early prophylactic introduction of low dose AED therapy (LEV or PER) in patients with moderate to severe middle cerebral artery infarct, could prevent the development of post-stroke epilepsy (primary prevention).

DETAILED DESCRIPTION:
Advance in stroke treatment have resulted in a dramatic reduction in the stroke mortality, however, the number of stroke survivors living with morbidity has increased significantly. Among the morbidities, seizures and epilepsy are not uncommon and post-stroke epilepsy has been identified as a significant clinical issue in stroke survivors. As we know, stroke is the most common cause of epilepsy in older adults and for patients aged more than 65, post-stroke epilepsy accounts for 30-50% of new-onset seizures (Tanaka and Ihara, 2017). The incidence of early seizures (occurring within the first 1-2 weeks of stroke) is between 2.4-5.4% and the risk of post-stroke late seizures (seizures occur later than 14 days of stroke) is around 7-18% (Shetty, 2013; Tanaka and Ihara, 2017). The stroke severity, location and type of pathological changes, genetic factors and pre-injury and post-injury exposure to non-genetic factors such as exposome can divide patients with ischemic stroke into different susceptibility (Pitkanen et al., 2016) and the standardized morbidity rate of developing epilepsy is highest during the first year. Our previous study also documented seizures during stroke presentation and during hospitalization would worsen the overall morbidity and mortality (Huang et al., 2014), suggesting the importance of awareness in seizure care in acute ischemic stroke. In addition, studies showed higher National Institutes of Health Stroke Scale (NIHSS) score, cortical involvement younger age, central nervous system (CNS) morbidities are associated with higher risk of post-stroke epilepsy (Tanaka and Ihara, 2017).

Occurrence of post-stroke epileptic seizure would lead to long-term poor prognosis and increased mortality (Bladin et al., 2000; Labovitz et al., 2001), and the post-stroke epilepsy has a high recurrence rate (Tanaka et al., 2017), which might lead to anxiety and worsen quality of life in the stroke survivors. As current treatments only focus on anti-seizure/anti-convulsion, based on our understanding of the epileptogenesis, we aim to develop a potential prophylactic treatment on patients with acute severe stroke to prevent from late occurrence of seizures and epilepsy.

Process of epileptogenesis is classically thought to occur in three phases: first the occurrence of a precipitating injury or event; second, a 'latent' period during which changes set in motion by the preceding injury act to transform the previously normal brain into an epileptic brain; and third, chronic, established epilepsy. It is during the latent period that the process of acquired epileptogenesis is thought to coalesce, and it is at this point in the process that interventions might be used to prevent the subsequent development of epilepsy (Goldberg and Coulter, 2013; Kikuyama et al., 2017). We have previously done researches on the medications that might have potential of anti-epileptogenesis in pilocarpine-induced animal models, supporting the concept of anti-epileptogenesis, giving intervention immediately following a brain insult (Lai et al., 2018, Hung et al., 2019).

Potential medications with potential of anti-epileptogenesis Based on our clinical experience, and laboratory researches (Huang et al., 2009, 2013; Lai et al., 2018; Hung et al., 2019), we have noted two newer AEDs with potential of anti-epileptogenesis. LEV, a current standard AED with a distinct synaptic vesicle modulating mechanism, has been demonstrated its potential in ameliorating epileptogenesis (Itoh et al., 2016; Kikuyama et al., 2017). Synaptic vesicle 2A (SV2A) is considered to play an important role for synaptic vesicle recycling and neurotransmitter excretion to the synaptic cleft, because mice lacking SV2A failed to grow, experienced severe seizures, and died within 3 weeks (Crowder et al., 1999). A clear correlation was seen between the affinity of LEV and its analogues to SV2A and the potency of their antiseizure protection in the mouse audiogenic model of epilepsy (Lynch et al., 2004). Furthermore, the LEV-treated adult male Node epileptic rats showed a significant increase of Bax/Bcl-2 mRNA expression ratio in the prefrontal cortex than the control group, but no change in the Bax/Bcl-2 mRNA expression ratio in hippocampus, suggesting the mechanism of acquired anti-epileptogenesis by LEV may be similar to spontaneous recovery of idiopathic generalized epilepsy during adolescence (Kikuyama et al., 2017). Our earlier study suggests its broad spectrum of modulating neuronal excitability (Huang et al., 2009). It is not metabolized through the P-450 hepatic cytochrome system and has not clinically relevant drug-drug interactions (Rosati et al., 2010). It has also been suggested as a first-choice drug against post-stroke seizures, based on safety and efficacy profiles in clinical studies (Belcastro et al., 2008). Thus, it is potentially worth investigation in primary prevention for patients with acute major stroke.

Perampanel (PER), a current standard antiepileptic drug with a distinct mechanism of selective non-competitive antagonist of alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA)-type receptors, has also been demonstrated its efficacy in treatment wide-spectrum epileptic seizures with good tolerability profile (Tyrlikova et al., 2008). Based on its block of glutamate excitotoxicity, PER is theoretically capable of modulating epileptogenesis and it has been demonstrated its potential in ameliorating epileptogenesis (Mohammad et al., 2019; Dupuis et al., 2017). As we know, the AMPA receptor has become a therapeutic target due to its involvement in ictogenesis and epileptogenesis. GluA2 subunit plays a role in calcium permeability. Thereby, AMPA receptor-mediated calcium signaling increases affects brain excitability. Recent report indicated that perampanel can block both calcium permeable and calcium in permeable AMPA receptors (Barygin et al., 2016). Our recent study on PER pharmacology also revealed it, for the first time, could inhibit voltage-gated sodium channels, suggesting its broad-spectrum properties in modulating neuronal excitability (Lai et al., 2019). Thus, it is potentially justified to evaluate if early administration of PER in patients with acute major stroke as a prophylactic therapy could hamper the development of epileptogenesis and the later post-stroke epilepsy.

Purpose of our study We aim to investigate if early administration of AEDs with potential anti-epileptogenesis could prevent the development of post-stroke epilepsy (primary prevention).

References:

1. Barygin OI. Inhibition of calcium-permeable and calcium impermeable AMPA receptors by perampanel in rat brain neurons. Neurosci Lett 2016;633:146-151.
2. Belcastro V, Costa C, Galletti F, Autuori A, Pierguidi L, Pisani F, Calabresi P, Parnetti L. Levetiracetam in newly diagnosed late-onset post-stroke seizures: a prospective observational study. Epilepsy Res 2008;82:223-6.
3. Bladin CF, Alexandrov AV, Bellavance A, Bornstein N, Chambers B, Cote R, Lebrun L, Pirisi A, Norris JW. Seizures after stroke: a prospective multicenter study. Arch Neurol 2000;57:e1617-22.
4. Crowder KM, Gunther JM, Jones TA, et al. Abnormal neurotransmission in mice lacking synaptic vesicle protein 2A (SV2A). Proc Natl Acad Sci USA 1999;96:15268-73.
5. Dupuis N, Enderlin J, Thomas J, Desnous B, Dournaud P, Allorge D, Auvin S. Anti-ictogenic and antiepileptogenic properties of perampanel in mature and immature rats. Epilepsia 2017;58:1985-92.
6. Goldberg E, Coulter D. Mechanisms of epileptogenesis: a convergence on neural circuit dysfunction. Nat Rev Neurosci. 2013;14:337-49.
7. Huang CW, Cheng JT, Tsai JJ, Wu SN, Huang CC. Diabetic hyperglycemia aggravates seizures and status epilepticus-induced hippocampal damage. Neurotox Res 2009;15:71-81.
8. Huang CW, Tsai JJ, Huang CC, Wu SN. Experimental and simulation studies on the mechanisms of Levetiracetam-mediated inhibition of delayed-rectifier potassium current (Kv3.1): Contribution to the firing of action potentials. J Physiol Pharmacol 2009;60:37-47.
9. Huang CW, Lai MC, Cheng JT, Tsai JJ, Huang CC, Wu SN. Pregabalin attenuates excitotoxicity in diabetes. PLOS One 2013;8:e65154-60.
10. Huang CW, Saposnik G, Fang J, Steven DA, Burneo JG. Influence of seizures on stroke outcomes: a large multicenter study. Neurology 2014;82:768-76.
11. Hung TY, Chu FL, Wu DC, Wu SN, Huang CW. The protective role of peroxisome proliferator-activated receptor-gamma in seizure and neuronal excitotoxicity. Mol Neurobiol 2019;56:5497-506.
12. Ikeda K, Sawada M, Morioka H, Kyuzen M, Ebina J, Nagasawa J, Yanagihashi M, Miura K, Ishikawa Y, Hirayama T, Takazawa T, Kano O, Kawabe K, Iwasaki Y. Clinical Profile and Changes of Serum Lipid Levels in Epileptic Patients after Cerebral Infarction. J Stroke Cerebrovasc Dis 2017;26:644-9.
13. Itoh K, Ishihara Y, Komori R. Levetiracetam treatment influences blood-brain barrier failure associated with angiogenesis and inflammatory responses in the acute phase of epileptogenesis in post-status epilepticus mice. Brain Res 2016;1652:1-13.
14. Kikuyama H, Hanaoka T, Kanazawa T, Yoshida Y, Mizuno T, Toyoda H, Yoneda H. The Mechanism of Anti-Epileptogenesis by Levetiracetam Treatment is Similar to the Spontaneous Recovery of Idiopathic Generalized Epilepsy during Adolescence. Psychiatry Investig 2017;14:844-50.
15. Labovitz DL, Hauser WA, Sacco RL. Prevalence and predictors of early seizure and status epilepticus after first stroke. Neurology 2001;57:200-6.
16. Lai MC, Hung TY, Lin KM, Sung PS, Wu SJ, Yang CS, Wu YJ, Jsai JJ, Wu SN, Huang CW. Sodium Metabisulfite: Effects on Ionic Currents and Excitotoxicity. Neurotox Res 2018;34:1-15.
17. Lai MC, Lin KM, Yeh PS, Wu SN, Huang CW. The novel effect of immunomodulator-glatiramer acetate on epileptogenesis and epileptic seizures. Cell Physiol Biochem 2018;50:150-68.
18. Lai MC, Tzeng RC, Huang CW, Wu SN. The Novel Direct Modulatory Effects of Perampanel, an Antagonist of AMPA Receptors, on Voltage-Gated Sodium and M-type Potassium Currents. Biomolecules 2019;9 pii: E638.
19. Lynch BA, Lambeng N, Nocka K, et al. The synaptic vesicle protein SV2A is the binding site for the antiepileptic drug levetiracetam. Proc Natl Acad Sci U S A 2004;101:9861-6.
20. Mohammad H, Sekar S, Wei Z, Moien-Afshari F, Taghibiglou C. Perampanel but Not Amantadine Prevents Behavioral Alterations and Epileptogenesis in Pilocarpine Rat Model of Status Epilepticus. Mol Neurobiol 2019;56:2508-23.
21. Morgenstern LB, Hemphill JC 3rd, Anderson C, Becker K, Broderick JP, Connolly ES Jr, Greenberg SM, Huang JN, Macdonald RL, Messe SR, Mitchell PH, Selim M, Tamargo RJ. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage. A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2010;41:2108-29.
22. Pitkanen A, Schwartzkroin PA, Moshe SM. Models of seizures and epilepsy. Burlington: Elsevier Academic Press. 2006.
23. Pitkanen A, Roivainen R, Lukasiuk K. Development of epilepsy after ischemic stroke. Lancet Neurol 2016;15:185-97.
24. Rosati A, Buttolo L, Stefini R. Efficacy and safety of levetiracetam in patients with glioma. Arch Neurol 2010;67:343-6.
25. Shetty A. Prospects of levetiracetam as a neuroprotective drug against status epilepticus, traumatic brain injury, and stroke. Front Neurol 2013;4:1-6.
26. Tanaka T, Ihara M. Post-stroke epilepsy. Neurochem Int 2017;107:219-28.
27. Tyrlikova I, Brazdil M, Rektor I, Tyrlik M. Perampanel as monotherapy and adjunctive therapy for focal onset seizures, focal to bilateral tonic-clonic seizures and as adjunctive therapy of generalized onset tonic-clonic seizures. Expert Rev Neurother 2018;18:1-12.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute MCA infarct (NIHSS > 8) and confirmed by brain MRI studies (excluding lacunar infarct) during hospital admission

Exclusion Criteria:

* Patients with prior clinical history of major stroke, significant head injury, brain tumor, major psychiatric illness, progressive neurodegenerative disorder, CNS infection, epilepsy, which might be precipitating to seizures or history of use of AEDs, including LEV or PER, during pregnancy or lactation, history of inadequate medical compliance, or any other significant major systemic disease with safety concern, determined by physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
post-stroke epileptic seizure | at least 14 days after stroke
  Occurrence of epileptic seizure following acute stage of stroke

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Wei Huang, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Chen YS, Sung PS, Lai MC, Huang CW. The Primary Prevention of Poststroke Epilepsy in Patients With Middle Cerebral Artery Infarct: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 24;12:e49412. doi: 10.2196/49412. PMID 37999939